CLINICAL TRIAL: NCT01974037
Title: Effects of Capsaicin on Salty Gustatory Cortices in Human
Brief Title: Capsaicin on Salty Gustatory Cortices
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhiming Zhu (Other)
Responsible Party: Sponsor-Investigator, Zhiming Zhu, Director of the Dept. of Hypertension & Endocrinology, Third Military Medical University
Organization: Third Military Medical University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: SATIETY-2
Record Dates: First submitted 2013-10-27; First posted 2013-11-01 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Volunteers
MeSH Terms: interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Capsaicin_effect subgroup 1 (Active Comparator): The volunteers allocated to the arm will perform neuroimaging detection with buccal administration of water with capsaicin.
  Interventions: Dietary Supplement: Capsaicin
- Capsaicin_effect subgroup 2 (Experimental): The volunteers allocated to the arm will perform neuroimaging detection with buccal administration of 100 mmol/L NaCl with capsaicin.
  Interventions: Dietary Supplement: Capsaicin
- Capsaicin_effect subgroup 3 (Experimental): The volunteers allocated to the arm will perform neuroimaging detection with buccal administration of 150 mmol/L NaCl with capsaicin.
  Interventions: Dietary Supplement: Capsaicin
- Capsaicin_effect subgroup 4 (No Intervention): The volunteers allocated to the arm will perform neuroimaging detection with buccal administration of 200 mmol/L NaCl.
- Salt_effect subgroup 1 (No Intervention): The volunteers allocated to the arm will perform neuroimaging detection with buccal administration of water.
- Salt_effect subgroup 2 (Experimental): The volunteers allocated to the arm will perform neuroimaging detection with buccal administration of 100 mmol/L NaCl.
  Interventions: Dietary Supplement: NaCl
- Salt_effect subgroup 3 (Experimental): The volunteers allocated to the arm will perform neuroimaging detection with buccal administration of 150 mmol/L NaCl.
  Interventions: Dietary Supplement: NaCl
- Salt_effect subgroup 4 (Experimental): The volunteers allocated to the arm will perform neuroimaging detection with buccal administration of 200 mmol/L NaCl.
  Interventions: Dietary Supplement: NaCl

INTERVENTIONS:
Dietary Supplement: Capsaicin — Capsaicin in the concentration of 0.5 µmol/L was mixed in the test solutions in Capsaicin_effect subgroups
  Arms: Capsaicin_effect subgroup 1; Capsaicin_effect subgroup 2; Capsaicin_effect subgroup 3
Dietary Supplement: NaCl — NaCl in various concentrations was desorved in the test solutions in Salt_effect subgroups
  Arms: Salt_effect subgroup 2; Salt_effect subgroup 3; Salt_effect subgroup 4

SUMMARY:
Excess dietary salt intake is closely associated with the development of hypertension and cardiocerebral vascular diseases. Preference of high salt diet might involve salty gustatory cortices change. This study focuses on examining the neuroimaging changes of salty gustatory cortices under different concentration of NaCl solution with or without capsaicin intervention through brain PET/CT scan.

DETAILED DESCRIPTION:
Hypertension and its related complications are common health problems that can lead to multiple organ damage and death. Excessive salt intake plays an important role in the development of hypertension.

The experimental design is a randomized, double-blind, interventional study to investigate the neuroimaging changes of salty gustatory cortices under different concentration of NaCl solution with or without capsaicin intervention through brain PET/CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 65 years.
* Willing and able to provide written informed consent.
* Willing and able to comply with all study procedures.

Exclusion Criteria:

* High basic metabolic rate, tumor, epilepsia.
* Hypogeusia or loss due to neural system disease or oral and digestive disease.
* Capsaicin allergy and poor compliance.
* Recently oral diuretics and participate in other pharmacological experiment in 3 months.
* Acute infection, cancer, serious arrhythmias, drug or alcohol abuse.
* Currently have cold, fever, acidosis, dehydration, diarrhea, vomiting during the study.
* Unwilling or unable to communication due to the dysnoesia and language disorders.
* Severe neural or psychiatric diseases that would preclude fully understand and corporation in the study.
* History of allergic reaction attributed to 18F-FDG.
* Pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Neuroimaging changes of salty gustatory cortices | 45min
  Buccal administration of test solution for five mins, and PET/CT scan after 40 mins

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, The Third Military Medical University, Chongqing, Chongqing Municipality, China